CLINICAL TRIAL: NCT03201653
Title: A Prospective Randomized Trial of Efficacy of Stump Closure for Distal Pancreatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201507019RIND
Record Dates: First submitted 2016-06-21; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2016-06

CONDITIONS: Pancreatic Fistula
Keywords: Distal Pancreatectomy; Pancreatic Fistula; Oxidized Regenerated Cellulose; Pancreatectomy
MeSH Terms: conditions — Pancreatic Fistula | interventions — Surgicel

STUDY DESIGN:
Intervention Model Description: SURGICEL group comparisons to traditional group (each performed at a nominal alpha of 0.05 and power of 0.80) in a 2:1 allocation ratio
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Stump closure as our institute routine, using interrupted silk mattress suture and continuous prolene sutures.
  Interventions: Procedure: Stump closure using NU-KNIT SURGICEL
- Surgicel (Experimental): Stump closure modified from our institute routine, using interrupted silk mattress suture and continuous prolene sutures with NU-KNIT SURGICEL overlying for reinforcement.
  Interventions: Procedure: Stump closure using NU-KNIT SURGICEL

INTERVENTIONS:
Procedure: Stump closure using NU-KNIT SURGICEL — We would use the Oxidized Regenerated Cellulose as NU-KNIT SURGICEL.
  Other Names: SURGICEL (Oxidized Regenerated Cellulose)

SUMMARY:
Overall morbidity rate remained high after distal pancreatectomy (DP), ranging from 30% to 60%. Whilst postoperative pancreatic fistula (POPF) remains serious and also is one of the most common complications after DP (12% to 40%). POPF after DP is also associated with major complications such as bleeding or septic shock and remains an equivocal problem. However, all the previous reports were retrospective review, non-randomized study, or individual experience and showed no significant improvement of overall POPF. As always, this issue remains in obscurity and seek for a more concrete evidence to solve.

DETAILED DESCRIPTION:
Pancreatic surgery has been called formidable operation not only the technical challenge to surgeons but also demanding for patients. It evolved into a safe procedure with mortality rates of <5% recently, cutting down gradually from 25% in the 1960s. However, overall morbidity rate remained high ranging from 30% to 60%.

Distal pancreatectomy (DP) has been believed a safer and minor procedure compared with pancreatic head resection including standard pancreaticoduodenectomy (PD), pylorus-preserving pancreaticoduodenectomy (PPPD), or duodenum-preserving pancreatic head resection (DPPHR). Whilst postoperative pancreatic fistula (POPF) remains serious and also is one of the most common complications after DP. Büchler et al observed that the POPF rate was in fact significantly higher after DP when compared to pancreatic head resections. The variable documented incidence of POPF following DP ranges from 12% to 40%. POPF after DP is also associated with major complications such as bleeding or septic shock and remains an equivocal problem.

Although the majority of complications are not life-threatening, POPF could prolong hospitalization, expend expenditure for healthcare, abrade the quality of life; moreover, delay in further management for a fraction of patients with malignancy. Over the past two decades, various risk factors and multitudinous operative procedures have been held for reduction POPD following DP. These include underlying disease process, method of stump closure, and concomitant splenectomy However, all these reports were retrospective review, non-randomized study, or individual experience. As always, this issue remains in obscurity and seek for a more concrete evidence to solve.

ELIGIBILITY:
Inclusion Criteria:

* age>= 20 years
* scheduled distal pancreatectomy at NTUH
* unable to realize this trial and willing to sign the informed consent form

Exclusion Criteria:

* age< 20 years, pregnent women, breast-feeding women, or mentally illed
* active malignancy within 2 years
* received other upper abdomen major surgery
* scheduled spleen preservation or associated major organ resection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
POPF rate | through study completion, an average of 16 days
  The percentage of overall (grade A, B, C) POPF.

SECONDARY OUTCOMES:
Duration of drainage replacement | through study completion, an average of 16 days
  Duration of drainage replacement after DP
Hospitalization | through study completion, an average of 16 days
  Duration of hospital stay after DP
Hospitalization cost | through study completion, an average of 16 days
  Total hospital cost of for DP
Mortality | 90 days
  Procedure-related mortality after DP

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No